CLINICAL TRIAL: NCT02233062
Title: Impact of Exclusive Enteral Nutrition Therapy on Sperm Quality of Male Patients With Crohn's Disease
Brief Title: Impact of Exclusive Enteral Nutrition Therapy on Sperm Quality of Patients With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Vice president, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140901; NSFC (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2014-09-01; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; semen quality; enteral nutrition; CDAI score higher than 150
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semen quality (Experimental)
  Interventions: Dietary Supplement: Exclusive Enteral Nutrition Therapy

INTERVENTIONS:
Dietary Supplement: Exclusive Enteral Nutrition Therapy

SUMMARY:
The purpose of this study is to investigate the impact of enteral nutrition therapy on sperm quality of patients with crohn's disease.

DETAILED DESCRIPTION:
The highest age- and sex-adjusted incidence rates for Crohn's Disease (CD) occur during the peak reproductive years. In addition, gastroenterologists frequently advise and manage patients with CD who desire to conceive. Enteral nutrition therapy is effective for induction and maintenance of remission in reproductive age men with CD. However, there is no available data on the effects of enteral nutrition therapy on semen quality. The purpose of this study is to investigate the impact of enteral nutrition therapy on sperm quality of patients with CD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn' Disease
* Male patients
* Age: 18-40 years old
* Receive 3-months exclusive enteral nutrition therapy

Exclusion Criteria:

* Used any experimental therapy in the 8 weeks before study entry date
* Had previously documented problems with male reproductive health, such as low sperm count, impotence, or malignancy
* The use of concomitant medication including sulphasalazine, 5-aminosalicylic acid or other immune-suppressives.
* Unable to complete the 3-months exclusive enteral nutrition therapy.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sperm motility | Up to 3 months
  Sperm motility is a useful marker of sperm quality. The normal level of sperm motility (World Health Organization criteria) should be higher than 50%.

SECONDARY OUTCOMES:
Crohn's Disease Activity Index | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling Hospital, Nanjing, Jiangsu, China